CLINICAL TRIAL: NCT07196514
Title: Exploring the Effects of an 8-week Turmeric Supplementation on Aspects of Physiology and Wellbeing in Healthy Older Adults
Brief Title: Effects of 8 Weeks of Turmeric Ingestion on Physiology and Wellbeing in Healthy Older Adults
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Nottingham Trent University (Other)
Collaborators: Innate-Essence Limited (Unknown)
Responsible Party: Principal Investigator, John Hough, Associate Professor in Health and Immunology, Nottingham Trent University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: 2268061
Record Dates: First submitted 2025-09-19; First posted 2025-09-29 (Actual); Last update posted 2026-01-16 (Actual); Status verified 2026-01

CONDITIONS: Turmeric; Placebo

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Placebo (Placebo Comparator): This group will take one placebo shot (containing a small amount of turmeric for taste-matching purposes) twice per day for 8 weeks.
  Interventions: Other: Placebo
- Turmeric (Experimental): This group will take one 60 mL commercially-available shot (containing 30% turmeric) twice per day for 8 weeks.
  Interventions: Dietary Supplement: Raw turmeric shots

INTERVENTIONS:
Dietary Supplement: Raw turmeric shots — This group will take one 60 mL commercially-available shot (containing 30% turmeric) twice per day for 8 weeks.
  Arms: Turmeric
Other: Placebo — This group will take one placebo shot (containing a small amount of turmeric for taste-matching purposes) twice per day for 8 weeks.
  Arms: Placebo

SUMMARY:
Curcumin (a bioactive compound found in turmeric) has demonstrated anti-inflammatory and antioxidant properties, and there is evidence to suggest that it may produce improvements in quality of life and markers of health in humans with various conditions. To date, the research has often focussed on the effects of curcumin in human participants with a particular condition. However, turmeric contains hundreds of other bioactive compounds (including other curcuminoids and essential oils) and may be able to benefit a wide range of older adults. Therefore, the aim of this study is to investigate the effects of twice daily consumption of a turmeric beverage for 8-weeks on the physiology and wellbeing of older adults (versus placebo).

ELIGIBILITY:
Inclusion Criteria:

- Body Mass Index between 18.5-39.9.

Exclusion Criteria:

* History of, or currently diagnosed with, a cardiovascular disease.
* Diagnosed with diabetes.
* Diagnosed with a liver, lung, or kidney disease.
* Diagnosed with osteoporosis.
* Diagnosed with dementia.
* Diagnosed with cancer.
* Use of medications/supplements/herbal remedies with human evidence of a significant interaction with turmeric.
* Allergy to turmeric, lemon, black pepper, watermelon, water, pineapple, magnesium or vitamin C.
* Pregnant, attempting to become pregnant, or breastfeeding.
* Regular (once per week or more) use of turmeric shots / supplements within the last 3 months.

Ages: 40 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2025-10-06 (Actual); Primary Completion 2026-07 (Estimated); Study Completion 2026-07 (Estimated)

PRIMARY OUTCOMES:
Plasma/serum Brain-derived neurotrophic factor | Two timepoints: 1) baseline 2) after 8 week intervention
  Measured using ELISA. We will analyse raw and percentage change values.
Plasma/serum total cholesterol | Two timepoints: 1) baseline 2) after 8 week intervention
  Measured using pentra C400 clinical chemistry analyser, We will analyse raw and percentage change values.
Chalder Fatigue Scale (CFS) | Two timepoints: 1) baseline 2) after 8 week intervention
  This questionnaire measures participants' severity of physical and mental fatigue. This will be scored "Likert style" from 0-33. Higher scores indicate greater levels of fatigue.

SECONDARY OUTCOMES:
Plasma/serum creatinine | Two timepoints: 1) baseline 2) after 8 week intervention
  Measured using pentra C400 clinical chemistry analyser, We will analyse raw and percentage change values.
Depression Anxiety Stress Scales - 21 items (DASS-21) | Two timepoints: 1) baseline 2) after 8 week intervention
  Participants choose from a range of questions designed to measure the severity of a range of symptoms common to both depression and anxiety. Scoring is based on a likert scale where higher scores relate to increased severity of depression, anxiety and stress.
McGill Pain Questionnaire | Two timepoints: 1) baseline 2) after 8 week intervention
  This questionnaire is used to evaluate a person experiencing significant pain. It can be used to monitor pain over time. Someone experiencing no pain would score 0 while the maximum score for pain would be 78.
36-Item Short Form Survey (SF-36) | Two timepoints: 1) baseline 2) after 8 week intervention
  This survey consists of generic questions covering eight health domains: physical functioning, bodily pain, role limitations due to physical health problems, role limitations due to personal or emotional problems, emotional well-being, social functioning, energy/fatigue, and general health perceptions. To score the survey, firstly, responses to items relate to scores between 0-100. Secondly, using a table, items in the same scale are averaged together to create the eight domains.
Plasma/serum ALT | Two timepoints: 1) baseline 2) after 8 week intervention
  Measured using pentra C400 clinical chemistry analyser, We will analyse raw and percentage change values.
Plasma/serum AST | Two timepoints: 1) baseline 2) after 8 week intervention
  Measured using pentra C400 clinical chemistry analyser, We will analyse raw and percentage change values.
Plasma/serum LDL cholesterol | Two timepoints: 1) baseline 2) after 8 week intervention
  Measured using pentra C400 clinical chemistry analyser, We will analyse raw and percentage change values.
Plasma/serum HDL cholesterol | Two timepoints: 1) baseline 2) after 8 week intervention
  Measured using pentra C400 clinical chemistry analyser, We will analyse raw and percentage change values.
Plasma/serum ALP | Two timepoints: 1) baseline 2) after 8 week intervention
  Measured using pentra C400 clinical chemistry analyser, We will analyse raw and percentage change values.
Serum GGT | Two timepoints: 1) baseline 2) after 8 week intervention
  Measured using pentra C400 clinical chemistry analyser, We will analyse raw and percentage change values.
Plasma/serum LDH | Two timepoints: 1) baseline 2) after 8 week intervention
  Measured using pentra C400 clinical chemistry analyser, We will analyse raw and percentage change values.
Plasma/serum creatine kinase | Two timepoints: 1) baseline 2) after 8 week intervention
  Measured using pentra C400 clinical chemistry analyser, We will analyse raw and percentage change values.
Plasma/serum C-reactive protein | Two timepoints: 1) baseline 2) after 8 week intervention
  Measured using pentra C400 clinical chemistry analyser, We will analyse raw and percentage change values.
Plasma/serum triglycerides | Two timepoints: 1) baseline 2) after 8 week intervention
  Measured using pentra C400 clinical chemistry analyser, We will analyse raw and percentage change values
Plasma/serum glucose | Two timepoints: 1) baseline 2) after 8 week intervention
  Measured using pentra C400 clinical chemistry analyser, We will analyse raw and percentage change values
Blood pressure | Two timepoints: 1) baseline 2) after 8 week intervention
  Systolic and diastolic blood pressure will be determined using an automatic upper arm blood pressure monitor. We will analyse raw and percentage change values.
Body mass | Two timepoints: 1) baseline 2) after 8 week intervention
  Determined by weighing participants.
Pittsburgh Sleep Quality Index (PSQI) | Two timepoints: 1) baseline 2) after 8 week intervention
  The PSQI is a tool used for assessing quality and disturbances over a one-month period. The sum of scores for the following 7 components, subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, use of sleeping medication and daytime function, are used to calculate a global PSQI score with scores greater than 5 indicating poor sleep quality.
N-back task for working memory (cognitive function) | Two timepoints: 1) baseline 2) after 8 week intervention
  This particular N-back tast comprises of only the 2-Back memory load. The total stimulus set is 15. Participants respond using the space bar when they see a stimulus that is presented two steps previously. There are three blocks consisting of 25 trials. Each stimulus will be presented for 500 ms and get 3 seconds to respond unless the participant responds earlier in which case the next trial will begin. Errors, correct responses, misses and reaction time, will be used as indices of performance. Commission errors or 'false alarms' occur when participants respond to non-targets.
Corsi forward block test for visuospatial working memory (cognitive function) | Two timepoints: 1) baseline 2) after 8 week intervention
  Participants are shown squares/blocks that light up one-by-one in a random order starting in a sequence length of two blocks. Participants then click with the mouse the blocks in exactly the same order as shown before. One extra square is added to each successfully completed sequence. If the participant fails to click the correct sequence they get one more chance with a different pattern and same sequence length. If they get it wrong again, the test ends and their score is shown (the corsi block span).
Corsi backward block test for visuospatial working memory (cognitive function) | Two timepoints: 1) baseline 2) after 8 week intervention
  This test is the reverse of the forward version. Participants are shown squares/blocks that light up one-by-one in a random order starting in a sequence length of two blocks. Participants then click with the mouse the blocks in the reverse order as shown before. One extra square is added to each successfully completed sequence. If the participant fails to click the correct sequence, they get one more chance with a different pattern and same sequence length. If they get it wrong again, the test ends and their score in shown (the corsi block span).
Sit-to-Stand Test | Two timepoints: 1) baseline 2) after 8 week intervention
  The objective of this test is to complete as many sit-to-stand repetitions as possible in 30 seconds. Participants will be instructed to sit in the middle of a chair placed against the wall with a seat height of 43 cm. Participants start with their feet flat on the floor, arms crossed at the wrists and held against the chest. On the signal, participants will rise to a full stand and return back to a fully seated position (counting as one full repetition). Before the test, participants will be allowed to practice 1-2 times to familiarise themselves with the movement
Hand Grip Strength Test | Two timepoints: 1) baseline 2) after 8 week intervention
  Participants will start by holding a hand grip dynamometer with their arm at a right angle and the elbow should be by the side of the body. The grip length will be noted and kept the same post intervention laboratory visit. Once the participant has a comfortable grip on the dynamometer they will squeeze the dynamometer with maximum isometric effort and maintain it for at least 5 seconds. No other body movement is allowed. The value shown on the dynamometer in kilograms will be recorded. Participants will alternate hands attempting the test three times with each hand.
2-minute Step Test | Two timepoints: 1) baseline 2) after 8 week intervention
  The objective of this test is to complete as many steps (with the knee reaching the marking) in 2-minutes as possible. To mark the line for the knee to cross, the distance between participant's anterior iliac crest and their patella will be measured and the midpoint will be found. A piece of tape will be placed on the stadiometer corresponding height of the midpoint between the patella and the iliac crest. The final score will be the number of times the right knee reached the tape height.
Waist circumference | Two timepoints: 1) baseline 2) after 8 week intervention
Waist to hip ratio | Two timepoints: 1) baseline 2) after 8 week intervention
Physical activity levels | Two one week periods: One week prior to intervention (baseline) and last week of intervention (week 8)
  A wrist monitor will allow for classifications of physical activity intensities (sedentary behaviour, light intensity physical activity, moderate intensity physical activity, moderate-vigorous intensity physical activity and vigorous intensity physical activity) and durations of time spent in these classifications.
Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) | Two timepoints: 1) baseline 2) after 8 week intervention
  Participants that have osteoarthritis will complete this questionnaire. The highest possible score is 96, which indicates the maximum pain, stiffness and difficulty with physical function.
Pain medication usage | Two timepoints: 1) Baseline 2) after 8 week intervention
  Pain medication usage over the prior 8 weeks will be assessed using a modified version of the Quantitative Analgesic Questionnaire.

CONTACTS AND LOCATIONS:
Locations (1):
- Nottingham Trent University, Clifton campus, Nottingham, United Kingdom

IPD SHARING:
Plan to Share IPD: No